CLINICAL TRIAL: NCT02488928
Title: E-PREDICT Evaluating the Predictive Value of EBUS ELASTOGRAPHY STRAIN in Patients With (Suspected) Lung Cancer
Brief Title: E- Predict: EBUS ELASTOGRAPHY STRAIN in Lung Cancer
Acronym: E-PREDICT
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-1676
Record Dates: First submitted 2015-06-19; First posted 2015-07-02 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2018-05

CONDITIONS: Lung Cancer
Keywords: NSCLC; EBUS; elastography; predictive value; strain
MeSH Terms: conditions — Lung Neoplasms; Sprains and Strains

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
EBUS elastography is a method to determine stiffness of lymph nodes, based on the minute deformation of the node by the beating heart. Whether EBUS elastography may further increase the sensitivity to predict the presence or absence of malignancy is unclear.

We suggest to use EBUS elastography strain pattern analysis for this assessment and correlate these measurements with the final pathology outcome to determine NPV, PPV, sensitivity and specificity of this analysis to predict the presence or absence of malignancy in patients with (suspected) lung cancer in a prospectively obtained observational cohort study.

DETAILED DESCRIPTION:
Patients will undergo a routine EBUS and/or EUS or EUSb with Pentax series EBUS or EUS scopes in combination with Hitachi Preirus Hi-Vision ultrasound processor with installed elastography software. Normal international guidelines for staging, diagnosis and specimen acquisition will be followed. For a normal evaluation B-mode measurements from all lymph node regions are obtained assessing size and standard ultrasound characteristics and all lymph nodes in the regions of interest that meet the criteria for fine needle aspiration will be sampled. For this study, in addition to the normal B-mode assessment of five sonographic B-mode characteristics elastography strain graph video, elastography image, and a strain histogram from the region of interest will be obtained.

Fine needle aspiration for cytology evaluation will be obtained from nodes based on imaging characteristics or standard sonography characteristics following current everyday clinical practice and the international guidelines. Subsequently, the patient charts will be retrospectively analysed after completion of the diagnostic and/or surgical treatment of the (suspected) lung cancer to match the obtained imaging data to pathology results (cytology and or histology where present) and clinical follow up until 6 months after the diagnostic procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for diagnostic or staging EBUS procedure for suspected or proven lung cancer.
* ASA physical status 1-3.
* Age 18 years or older.

Exclusion Criteria:

* Bleeding disorders.
* Contra-indication for temporary interruption of the use of anticoagulant therapy (acenocoumarol, warfarin, therapeutic dose of low molecular weight heparines or clopidrogel).
* Known allergy for lidocaine.
* Uncontrolled pulmonary hypertension.
* Recent and/or uncontrolled cardiac disease.
* Compromised upper airway (eg concomitant head and neck cancer or central airway stenosis for any reason).
* Prior radiotherapy treatment involving the central airways
* ASA classification greater than or equal to 4.
* Pregnancy.
* Inability to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or proven lung cancer are eligible if there is an indication for EBUS, EUS or combined EBUS and EUSb (single scope, EUS with EBUS scope). Eligible are patients with no contra-indications for EBUS.
Sampling Method: Non-Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
stiffness of lymph nodes | participants will be followed for the duration of hospital stay, an expected average of 4 hours
  stiffness/strain is a relative measure and has therefor no units

CONTACTS AND LOCATIONS:
Overall Officials: Erik van der Heijden, MD, PhD, Principal Investigator — chest physician
Locations (7):
- Rigshospitalet, Copenhagen, Denmark
- Italy (4):
  - Interventional Pulmonology Unit Policlinico S. Orsola-Malpighi, Bologna
  - Azienda Ospedaliera Universitaria di Careggi, Florence
  - Ausl Modena - Ospedale Santa Maria Bianca, Modena
  - Pesaro-Fano Hospital, Pesaro
- Netherlands (2):
  - RadboudUMC, Nijmegen, Gelderland
  - Academic Medical Center, Amsterdam